CLINICAL TRIAL: NCT05750862
Title: Accuracy of Topography Guided Automatic Marking of the Intraocular Lens (IOL) -Axis in Toric IOL-impantation in Femtosecond Laser Assisted Cataract Surgery (FLACS). A Prospective Non-randomised Controlled Study
Brief Title: Accuracy of Topography Guided Automatic Marking of the Intraocular Lens (IOL) -Axis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Frank Bochmann (Other)
Responsible Party: Sponsor-Investigator, Frank Bochmann, PD Dr. med., Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023_D0001
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cataract Senile; Astigmatism
Keywords: Cataract; Astigmatism; Toric intraocular lens alignment
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): Study with one single arm. All participants will receive two interventions that will be compared to each other.
  Interventions: Procedure: Marking of the intended axis of IOL-Implantation manually with an ink and marking device on the surface of the eye

INTERVENTIONS:
Procedure: Marking of the intended axis of IOL-Implantation manually with an ink and marking device on the surface of the eye — The marking of the intended implantation axis of the interocular lens will be marked in all patients with topography guided in the corneal stroma with laser and in addition manually with a caliper and ink on the corneal surface
  Other Names: Autotmated, topopgraphy guided marking of the inteded axis of IOL-Implantation with the Catalys femtosecond laser

SUMMARY:
In cataract surgery, the opaque lens is replaced by an artificial intraocular lens. The procedure also allows for correction of an refractive error such as myopia, hyperopia or astigmatism. In case of correction of an astigmatism, the axis intraocular lens has to be alligned to the axis of the corneal astigmatism. There are serveral options, the intendet position of the axis can be marked on the cornea, either manually using ink and a special caliper or with an automatic laser device.

The aim of this study is to assess the accuracy of topography guided automatic marking of the intended IOL-axis in toric IOL-implantation in femtosecond laser assisted cataract surgery (FLACS)

DETAILED DESCRIPTION:
In cataract surgery, the opaque lens is replaced by an artificial intraocular lens. Based on a preoperative measurement of the eye (biometry) the power of the artificial lens is calculated so that refractive errors may be corrected. If high corneal astigmatism is present a correction of this astigmatism is also possible and offered to the patients. This may lead to a certain degree of spectacle independence. The astigmatism is corrected by the implantation of a special toric lens (spherical and cylindrical correction). This toric lens has to be positioned in the eye so that the axis of the IOL-cylinder aligns 90° to the axis of the corneal cylinder. The axis of the corneal cylinder has to be measured and marked before the intervention. Usually, the intended axis of placement for the toric IOL is marked with ink at the slitlamp or with the aid of a manual axis instrument. Anatomical landmarks without preoperative marking are also used. A clinical trends survey of the European society of cataract and refractive surgery (ESCRS) for 2021 has revealed that in 15% of all cataract cases (totally 550'000 cases assessed) a special toric IOL was implanted to correct a clinically significant astigmatism. About 75% use manual marking with ink. Only 25% of cases were operated using a digital image registration.

The manual marking using a marking device is currently the gold standard. However, the manual marking might be not very precise. The thick ink-marks on the cornea and the limbus are not very well visible. Sometimes the marks are not perfectly centred on the optical axis of the eye. Head tilt and rotation of the eyeball if patients are not fixating may lead to a deviation up to several degrees.

One possible solution of this problem are digital imaging technologies. The Cassini topography instrument for example provides additional to the measurement of the axis and the cylindrical power of the cornea a digital image of the iris. If the cataract surgery is performed assisted by a femtosecond laser (FLACS), this digital image is transferred to the femtosecond laser. Based on this image the software of the laser is capable to determine the correct position of the axis of the cylinder of the cornea and the femtosecond laser can make two intrastromal marks in the cornea. These marks allow the surgeon to align the toric IOL without any preoperative manipulations with ink and marking tools.

The aim of this study is to assess the accuracy of topography guided automatic marking of the intended IOL-axis in toric IOL-implantation in femtosecond laser assisted cataract surgery (FLACS)

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cataract surgery who opt for a femtolaser-assisted cataract surgery (FLACS) and Implantation of a toric intraocular lens. (both are extra options not covered by the insurance)
* Corneal astigmatism more than 1.o diopters confirmed in a measurement of corneal topography (Pentacam and Cassini topography devices)

Exclusion Criteria:

* Earlier corneal or intraocular refractive interventions (C-TEN, Lasik…)
* Irregular corneal astigmatism
* Corneal pathologies associated with ectasia and/or irregular astigmatism (Pterygium, Keratoconus, pellucide marginal degeneration…)
* Earlier intraocular or ocular surface involving surgeries
* Severe dry eye disease
* Contraindication of performing cataract surgery under topical anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Deviation of laser marking | 1 month
  Deviation of laser marking in the cornea compared to intended position of the axis in degrees
Difference of laser marking | 1 month
  Difference of laser marking in the cornea compared to manual ink marking in degrees.

SECONDARY OUTCOMES:
Reduction of astigmatism | 1 month
  Total of reduction of astigmatism in the postoperative refraction
Decentration of manual ink marking | 1 month
  Decentration of the ink marking (yes or no)
correction of IOL position | 1 month
  Number of necessary corrections of IOL-position

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bochmann, MD, Principal Investigator — Eye Clinic, Cantonal Hospital of Lucerne, Switzerland
Locations (1):
- Eye Clinic, Cantonal Hospital of Lucerne, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
it is not foreseen to make individual participant data available to the researchers